CLINICAL TRIAL: NCT02697240
Title: A Phase 1 Dose Escalation Study of Continuous Intravenous L-citrulline During Sickle Cell Pain Crisis or Acute Chest Syndrome
Brief Title: A Phase 1 Study of Continuous Intravenous L-citrulline During Sickle Cell Pain Crisis or Acute Chest Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Suvankar Majumdar, Associate Professor, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0230
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; citrulline
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravenous citrulline (Experimental): Intravenous citrulline at a bolus dose over 5 minutes and then a continuous rate for the next 23 hours.
  Interventions: Drug: Intravenous citrulline

INTERVENTIONS:
Drug: Intravenous citrulline — Intravenous citrulline at a bolus dose of 20 mg/kg over 5 minutes and then continuous at a rate of 7 mg/kg/hour for the next 23 hours for the first 7 participants, and depending on safety and pharmacokinetic profile, increase or decrease the continuous rate to 9 or 5 mg/kg/hour for the next 7 participants.

SUMMARY:
Sickle cell disease is a genetic red blood cell disorder characterized by vaso-occlusion from sickling of red blood cells, that can lead to pain or organ complications such as acute chest syndrome. Sickle cell disease is associated with low amounts of nitric oxide, a compound important for dilating the blood vessel wall. Citrulline is a substance that is known to increase nitric oxide. The goal of this Phase I study are to find the highest safe dose of continuous IV citrulline that can be given to individuals with sickle cell disease experiencing a sickle cell pain crisis or acute chest syndrome without causing severe side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Sickle cell disease genotypes (HbSS, HbS/β0-thalassemia, HbS/β+-thalassemia, HbSC)
2. Ages 6 to 50 years old
3. Patients with sickle cell disease aged 6 to 50 years old Presence of sickle cell pain crisis defined by the presence of pain requiring hospitalization and parental opioid therapy
4. Presence of acute chest syndrome defined by the presence of a new CXR infiltrate and any one of the following respiratory symptoms of fever, shortness of breath, wheezing, chest pain, cough or new onset hypoxia.

Exclusion Criteria:

1. Presence of any other complication related to sickle cell disease requiring hospitalization such as splenic sequestration, hepatic sequestration, stroke, avascular necrosis of the hip/shoulder, acute priapism, etc.
2. Severe anemia (hemoglobin < 5g/dL)
3. History of red blood cell transfusion within the last 30 days
4. Systemic steroid therapy within the last 48 hours
5. Pregnant (as confirmed by a negative urine pregnancy test) or lactating female
6. Alanine/aspartate transferase >2x upper limit of normal laboratory range for age.
7. Subject has the following serum creatinine:

   * Age 6 to 13 years > 0.9 mg/dL
   * Age 14-17 years 1.0 mg/dL
   * Age 18 years >1.5mg/dL
8. Patients with an inability to give consent will be excluded

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2016-02; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barr FE, Tirona RG, Taylor MB, Rice G, Arnold J, Cunningham G, Smith HA, Campbell A, Canter JA, Christian KG, Drinkwater DC, Scholl F, Kavanaugh-McHugh A, Summar ML. Pharmacokinetics and safety of intravenously administered citrulline in children undergoing congenital heart surgery: potential therapy for postoperative pulmonary hypertension. J Thorac Cardiovasc Surg. 2007 Aug;134(2):319-26. doi: 10.1016/j.jtcvs.2007.02.043. PMID 17662768

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Citrulline
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intravenous Citrulline
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 19.5 [18 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The number and severity of adverse event will be determined according to the NCI Common Terminology Criteria for Adverse Events (CTCAE)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Citrulline
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Plasma Citrulline Level
Time Frame: Plasma citrulline levels will be evaluated at the following time points: trough level, 10 minutes (peak level), 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours and 48 hours, to evaluate the pharmacokinetic profile
Measure: Mean (Standard Deviation); unit: micromol/hr/kg
Arm/Group | Intravenous Citrulline
Number analyzed (Participants) | 4
micromol/hr/kg | 5 (2.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 4 weeks from study drug administration
Arm/Group | Intravenous Citrulline
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Citrulline (N=4)
transaminitis (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT02697240/Prot_SAP_000.pdf